CLINICAL TRIAL: NCT06073626
Title: Addressing Genomic Disparities in Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Georgetown University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anita Y. Kinney, PhD, RN, Director at Rutgers Cancer Institute, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Pro2022001513; R01CA277599 (NIH)
Record Dates: First submitted 2023-09-14; First posted 2023-10-10 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Hereditary Cancer; Genetic Testing
Keywords: hereditary cancer; genetic testing; genetic education; relational agent; chatbot

STUDY DESIGN:
Intervention Model Description: This study will employ a 2-arm parallel group randomized controlled trial to evaluate the efficacy of the relational agent/chatbot (RA) intervention compared to Enhanced Usual Care (EUC) among 428 Black cancer survivors. Randomization is at the patient level and will be balanced in a 1:1 ratio - with 214 participants randomized to each arm. Randomization will be in blocks and stratified by recruitment site (DC, NJ). The investigators also plan to enroll a total of 16 usability testing participants across all sites.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Treating clinicians will be blind their patients group assignment. While participants cannot be blinded to group, they will be blinded to the study's specific hypotheses. Statisticians and outcome assessors will be blinded to allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relational Agent (RA) (Experimental): Participants in the RA arm will receive a clinical letter from the institution's clinical genetics program with a link to the RA. The fully HIPAA-compliant RA will provide comparable educational information to traditional genetic counseling (GC) but in a streamlined and tailored manner including video, education and decision support, patient testimonial and answers to questions in real-time. Participants will be informed that they may speak to a genetic risk specialist free of charge. For participants who wish to proceed directly to GT, the RA will alert staff to these requests and a GT kit will be mailed to them. Results will be shared with the participant, their oncologist and tailored per the result. Participants who indicate that they are unsure or do not want GT will be encouraged by RA to discuss their risk and GT options with their oncology provider and to schedule a GC appointment with the clinic.
  Interventions: Behavioral: Relational agent (RA) / Chatbot
- Enhanced Usual Care (EUC) (Active Comparator): Participants in the EUC arm will also be mailed a clinical letter signed by the Medical Director of the institution's clinical genetics program. The letter sent to EUC participants will inform them of their own and their family's potential risk for carrying a pathogenic variant (PV) related to hereditary cancer. The letter will emphasize their eligibility for GT, include a recommendation to consider scheduling a GC appointment to obtain more information, and include a link to the Rutgers Cancer Institute or LCCC high-risk clinic website. The study team will help facilitate GT when requested by the participant. Results will be shared with the participant, their oncologist and tailored per the result.
  Interventions: Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: Relational agent (RA) / Chatbot — Consists of clinical letter and engagement with genetic education and uptake of genetic testing for hereditary cancer risk among Black cancer survivors.
  Arms: Relational Agent (RA)
Behavioral: Enhanced Usual Care (EUC) — Consists of clinical letter and recommendation for genetic testing for hereditary cancer risk among Black cancer survivors.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
The goal of this observational study is to increase genetic education and genetic testing for hereditary cancer risk among Black cancer survivors. The study will:

1. Test the effectiveness of a chatbot intervention (also called relational agent, or RA) vs. enhanced usual care (EUC) on engagement in genetic education and requests for genetic testing.
2. Evaluate the impact of the chatbot vs. EUC on the process that participants use to make decisions and evaluate effects on well-being (also called psychosocial outcomes).
3. Explore the ways (methods) that influence how participants experience the intervention.
4. Explore the feasibility of incorporating a Family Sharing Portal (FSP) for participants who receive a positive test result, to facilitate family communication of these test results and genetic testing of first-degree biological relatives after they have received genetic education by the RA.

The main questions this study aims to answer are which group - the chatbot (RA) group or the EUC group - is more likely to request genetic testing and which group is more likely to get (engage with) genetic education.

Participants will be randomly assigned to either the chatbot (RA) group or EUC group. This means each participant has an equal chance of being placed in either group, just like flipping a coin. Each group will receive genetic education and have an opportunity to request genetic testing. Researchers will compare the chatbot (RA) group and the EUC group to see which may request more GT (genetic testing) and which group engages more with genetic education.

DETAILED DESCRIPTION:
Research Design and Methods:

This study will employ a 2-arm parallel group randomized controlled trial to evaluate the efficacy of the RA intervention compared to EUC among 428 Black cancer survivors who meet the National Comprehensive Cancer Network's guidelines for genetic referral. Primary outcomes will be engagement with genetic education and uptake of genetic testing (Aim 1). The investigators will also evaluate the impact of the RA intervention on psychosocial and decision quality outcomes (Aim 2) and evaluate mediators and moderators of intervention impact (Aim 3). In response to patient identified needs, we will also explore the feasibility of incorporating a Family Sharing Portal (FSP). All participants who receive a positive test result will be input into the FSP (Aim 4).

Research Procedures:

The design for this study is a 2-arm parallel group trial. Randomization is at the patient level. The investigators will recruit eligible cancer survivors who will be randomized by computer to enhanced usual care (EUC) or RA. Randomization will be balanced in a 1:1 ratio - with 214 participants randomized to each arm. Because this study is designed to address the disparity of low genetic testing utilization in Black cancer patients, all study participants will be Black and approximately 10% will be Hispanic.

The investigators will utilize the EHRs at our participating sites to identify cancer survivors who have not been tested despite meeting GT eligibility criteria. Participants will be ascertained from 1) Georgetown Lombardi Comprehensive Cancer Center (LCCC), MedStar Washington Cancer Institute (MWCI) and MedStar Franklin Square Medical Center in DC and 2) Rutgers' Cancer Institute (in New Brunswick and at University Hospital Newark) including RWJ Barnabas Health community oncology sites. Participants will be women and men who self-identify as Black or African American, have a history of breast, ovarian, uterine, colorectal, prostate, or pancreatic cancer, are at least six-months post-diagnosis, and have received care at one of the participating sites in the prior five years. There is no limit on the years since diagnosis as genetic testing (GT) can guide treatment decisions and provide opportunities for cascade testing to guide screening and prevention in at-risk relatives.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* Self-identify as Black or African American
* At least 6-months post diagnosis with any of the following cancers: breast, ovarian, uterine, prostate, colorectal, pancreatic
* Have not had genetic testing for hereditary cancer
* Have received care at one of the participating sites in the prior five years
* Meet National Comprehensive Cancer Network criteria for germline GT
* Able to read and speak in English
* Capable of providing informed consent
* Have internet access (via smartphone, tablet or computer)
* Comfortable using a computer or mobile phone independently to access information

Exclusion Criteria:

* Do not speak English
* Unable to access the Internet
* Have previously undergone germline genetic testing for hereditary cancer risk or previously had genetic counseling (GC) and declined genetic testing (GT)
* Are unable to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Uptake of Germline Genetic Testing | 6-months
  As captured via internal RedCap form for the number or count of participants who opt for genetic testing, the investigators will test the efficacy of a culturally tailored and interactive electronic relational agent (RA) intervention vs. enhanced usual care (EUC) consisting of clinical letter and genetic recommendation on engagement in genetic testing uptake;
Survey Assessment of Impact of RA vs. EUC | 1-month and 6-month survey
  Evaluate the impact of the RA vs. EUC on informed decision-making and psychosocial outcomes via survey measures of related constructs at 1-month and 6-month surveys. Multiple scales are used to measure this outcome and each scale has a unique scoring system.
Survey Assessment of Mediators and Moderators of Efficacy | Baseline, 1-month and 6-month surveys
  Explore potential mechanisms by assessing mediators and moderators of efficacy via survey measures of related constructs at baseline, 1-month and 6-month surveys. Multiple scales are used to measure this outcome and each scale has a unique scoring system.

SECONDARY OUTCOMES:
Survey Assessment of Engagement with Genetic Education | 1-month survey
  Engagement with genetic education/counseling via survey measures of related constructs at 1-month survey. Multiple scales are used to measure this outcome and each scale has a unique scoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Y Kinney, PhD, RN, Principal Investigator — Director at Rutgers Cancer Institute
Locations (2):
- United States (2):
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Rutgers Cancer Institute, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] An J, Huq M, Speiser E, Grumet S, Peshkin BN, Heidt E, Adams-Campbell L, Grisham C, Tundealao S, Yesha R, Toppmeyer D, Isaacs C, Sorgen L, Tan N, Hooda-Nehra A, Nix MA, Reed DJ, Staton J, Schwartz MD, Kinney AY. Expanding access to cancer genetic care for cancer survivors: Rationale and design for a randomized controlled trial of a chatbot-based genetic education and testing. Contemp Clin Trials. 2026 Jan 17:108217. doi: 10.1016/j.cct.2026.108217. Online ahead of print. PMID 41554333